CLINICAL TRIAL: NCT00320424
Title: Clinical Evaluation of GSK576428 (Fondaparinux Sodium) in Prevention of Venous Thromboembolism After Hip Fracture Surgery
Brief Title: Hip Fracture Study of GSK576428 (Fondaparinux Sodium)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AR3106335
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Results first posted 2017-10-11 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Thromboembolism
Keywords: Xa factor; VTE; MOSLL; pentasaccharide
MeSH Terms: conditions — Thromboembolism | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Fondaparinux

SUMMARY:
This study is requested by PMDA to confirm the efficacy and the safety for HFS.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip fracture surgery within 10 days following the time of fracture of the hip (proximal femur) (or following the time of fracture estimated from trauma).

Exclusion Criteria:

* Active, clinically significant bleeding (excluding drainage).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-02-16 (Actual); Primary Completion 2006-10-26 (Actual); Study Completion 2006-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 48 participants undergoing major orthopedic surgery of the lower limb such as hip fracture surgery, knee replacement surgery and hip replacement surgery were enrolled from 16 February 2006 to 26 October 2006 at 9 centers in Japan. The safety population consisted of 48 participants and full analysis set consisted of 37 participants.
Groups:
- Fondaparinux Sodium 2.5 mg s.c.: Participants received fondaparinux sodium 2.5 milligrams (mg) by subcutaneous (s.c.) injection for 14 days between Day 2 to Day 11-15. The first injection of the study drug was given 24 ± 2 hours after surgical closure. From Day 3 onwards, the injection of the study drug was given at about the same time every day as far as possible (but more than 12 hours after the first dose on Day 2).
Period: Overall Study
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Started | 48
Completed | 42
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Groups:
- Fondaparinux Sodium 2.5 mg s.c.: Participants received fondaparinux sodium 2.5 mg by s.c. injection for 14 days between Day 2 to Day 11-15. The first injection of the study drug was given 24 ± 2 hours after surgical closure. From Day 3 onwards, the injection of the study drug was given at about the same time every day as far as possible (but more than 12 hours after the first dose on Day 2).
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 48

OUTCOME MEASURES:

1. Primary Outcome: Rate of Major Bleeding During Treatment Period
Description: Rate (%) was defined as number of events divided by the number of participants evaluated multiplied by 100. Signs and symptoms suggestive of venous thromboembolic events (VTE) included, but were not limited to lower extremity deep vein thrombosis (DVT): erythema, warmth, pain, swelling, tenderness and pulmonary embolism (PE): pleuritic chest pain, dyspnea, cough, hemoptysis, syncope, light-headedness/dizziness, tachypnea, and tachycardia. Intended treatment period started 24±2 hours after surgical closure. Venogram was obtained not later than 2 calendar days after the last study drug administration (between Day 11 and 17). These events were adjudicated by the Central Independent Adjudication Committee of Efficacy (CIACE).
Time Frame: From the first study drug injection up to Day 17
Population: Full analysis set used which consisted of all participants who were assigned to study drug with the exception of those who did not receive study drug at all and those with no valid efficacy data (example no evaluable venogram).
Measure: Number (95% Confidence Interval); unit: % of normalized events per participant
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 37
% of normalized events per participant | 21.6 [9.8 to 38.2]

2. Secondary Outcome: Rate of PE During Treatment Period
Description: Rate (%) was defined as number of events divided by the number of participants evaluated multiplied by 100. Signs and symptoms suggestive of VTE included, but were not limited to lower extremity PE: pleuritic chest pain, dyspnea, cough, hemoptysis, syncope, light-headedness/dizziness, tachypnea, and tachycardia. Intended treatment period started 24±2 hours after surgical closure. Venogram was obtained not later than 2 calendar days after the last study drug administration (between Day 11 and 17). These events were adjudicated by the CIACE. It was evaluated from the first study drug injection up to Day 17 or to first venogram, whichever occurred first.
Time Frame: Up to Day 17
Population: Safety population used which consisted of all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: % of normalized events per participant
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 48
% of normalized events per participant | 0 [0 to 0]

3. Secondary Outcome: Rate of DVT During Treatment Period
Description: Rate (%) was defined as number of events divided by the number of patients evaluated multiplied by 100. Signs and symptoms suggestive of VTE included, but were not limited to lower extremity DVT: erythema, warmth, pain, swelling, tenderness. Intended treatment period started 24±2 hours after surgical closure. Venogram was obtained not later than 2 calendar days after the last study drug administration (between Day 11 and 17). These events were adjudicated by the CIACE. It was evaluated from the first study drug injection up to Day 17 or to first venogram, whichever occurred first.
Time Frame: Up to Day 17
Population: Efficacy evaluable participants used consisted of a subpopulation of safety population who were judged to be evaluable for all DVT and proximal DVT or distal only DVT by the site of occurrence (total/side of operation/opposite side of operation/both sides). Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: % of normalized events per participant
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 37
% of normalized events per participant | 21.6

4. Secondary Outcome: Rate of Proximal DVT During Treatment Period
Description: Rate (%) was defined as number of events divided by the number of participants evaluated multiplied by 100. Signs and symptoms suggestive of VTE included, but were not limited to lower extremity DVT: erythema, warmth, pain, swelling, tenderness. Intended treatment period started 24±2 hours after surgical closure. Venogram was obtained not later than 2 calendar days after the last study drug administration (between Day 11 and 17). These events were adjudicated by the CIACE. It was evaluated from the first study drug injection up to Day 17 or to first venogram, whichever occurred first.
Time Frame: Up to Day 17
Population: Efficacy evaluable participants used. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: % of normalized events per participant
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 38
% of normalized events per participant | 2.6

5. Secondary Outcome: Rate of Distal Only DVT During Treatment Period
Description: as for outcome 4
Time Frame: Up to Day 17
Population: as for outcome 4
Measure: Number; unit: % of normalized events per participant
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 37
% of normalized events per participant | 21.6

6. Secondary Outcome: Number of Participants With Major Bleeding During Treatment Period
Description: Major bleeding events were defined as clinically unusual bleeding meeting any of the following criteria: fatal bleeding, bleeding including retroperitoneal and intracranial bleeding or bleeding into a critical organ (eye, adrenal gland, pericardium, spine), reoperation due to bleeding/hematoma at the operative site, bleeding leading to a hemoglobin (Hb) fall >=2 grams per deciliter (g/dL, 1.6 millimoles per liter [mmol/L]) within 48 hour of the bleed, bleeding that required a transfusion of red blood cell or whole blood derived from >=900 millilters (mL) of whole blood within 48 hours of the bleed (excluding the autologous transfusion except for the treatment of bleeding adverse event (AE) and bleeding leading to the bleeding index (BI) >=2. Major bleeding events were adjudicated by the Central Independent Adjudication Committee of Safety (CIACS).
Time Frame: From the first study drug injection up to 2 days after the last study drug injection (approximately up to Day 17)
Population: Safety population used.
Measure: Count of Participants; unit: Participants
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 48
Participants | 0

7. Secondary Outcome: Number of Participants With Minor Bleeding and Any Bleeding (Major and/or Minor Bleeding)
Description: Minor bleeding and any bleeding (major and/or minor bleeding) events were adjudicated by the CIACS. Minor bleeding was defined as clinically overt bleeding not meeting the criteria for major bleeding and considered more than expected in the clinical context. Any bleeding (major and/or minor bleeding) could be recorded may be major and/or minor.
Time Frame: From the first study drug injection up to 2 days after the last study drug injection (approximately up to Day 17)
Population: Safety population used.
Measure: Count of Participants; unit: Participants
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 48
Participants
  Minor Bleeding | 0
  Any Bleeding | 0

8. Secondary Outcome: Number of Participants With Adverse Events (AE), Serious Adverse Events (SAE) and Death
Description: An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Time Frame: From the first study drug injection up to 2 days after the last study drug injection (approximately up to Day 17)
Population: Safety population used.
Measure: Count of Participants; unit: Participants
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 48
Participants
  Any AE | 37
  Any SAE | 2
  Death | 0

9. Secondary Outcome: Number of Transfused Participants
Description: Blood product transfusions consisted of packed red blood cells or fresh frozen plasma or both. This was done between Day 2 and 2 calendar days after the last injection.
Time Frame: From the first study drug injection up to 2 days after the last study drug injection (approximately up to Day 17)
Population: Safety population used.
Measure: Count of Participants; unit: Participants
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 48
Participants | 1

10. Secondary Outcome: Summary of Units Transfused
Description: as for outcome 9
Time Frame: From the first study drug injection up to 2 days after the last study drug injection (approximately up to Day 17)
Population: Safety population used.
Measure: Number; unit: mL
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 48
mL | 280

11. Secondary Outcome: Rate of Symptomatic DVT
Description: as for outcome 4
Time Frame: Up to Day 17
Population: Safety population used.
Measure: Number; unit: % of normalized events per participant
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
Number analyzed (Participants) | 48
% of normalized events per participant | 0

ADVERSE EVENTS:
Time Frame: AE and SAE were reported throughout the study (from the first study drug injection up to 2 days after the last study drug injection [approximately up to Day 17]).
Description: Safety population was used for reporting AE and SAE.
Arm/Group | Fondaparinux Sodium 2.5 mg s.c.
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 2/48
Other Adverse Events (participants affected / at risk) | 37/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux Sodium 2.5 mg s.c. (N=48)
Ileus (Gastrointestinal disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux Sodium 2.5 mg s.c. (N=48)
Constipation (Gastrointestinal disorders) | 8
Insomnia (Psychiatric disorders) | 8
Oedema peripheral (General disorders) | 4
Excoriation (Injury, poisoning and procedural complications) | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4
Restlessness (Psychiatric disorders) | 3
Pyrexia (General disorders) | 3
Blood alkaline phosphatase increased (Investigations) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
C reactive protein increased (Investigations) | 2
Platelet count increased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Nasopharyngitis (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.